CLINICAL TRIAL: NCT00006513
Title: Assessing the Occupation Burden in COPD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 949; R01HL067438 (NIH)
Record Dates: First submitted 2000-11-20; First posted 2000-11-21 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2006-01

CONDITIONS: Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To assess the population burden of occupational exposures in the prevalence and progression of chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
BACKGROUND:

Chronic obstructive pulmonary disease is the only one of the top four or five leading causes of death in the U.S. with worsening epidemiological trends. Cigarette smoking accounts for approximately 85 percent-90 percent of cases, but the other 10 percent-15 percent of the attributable risk still represents a substantial fraction of this disease that remains unexplained. Recently, several studies, in various countries, have addressed whether certain occupational exposures (primarily those relating to dusts, vapors, gases, and/or fumes) are potential risk factors for COPD. Most of these studies have shown elevated odds ratios or relative risks, although not always to a statistically significant level.

DESIGN NARRATIVE:

A population sample of the continental United States of those aged 55-75, supplemented by an enriched sample in geographic "hot spots" identified by the National Institute for Occupational Safety and Health (NIOSH) through respiratory diseases mapping. Structured telephone interviews assessed demographics, health status, smoking exposures, and occupational histories. High risk jobs were coded using a job matrix system independent of subject report of specific exposures. Two hundred thirty-four of those with COPD, with over-sampling of those with greater severity, were followed at 12-14 months to assess health status and health services utilization, as well as decrements in quality of life.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Blanc — University of California, San Francisco

REFERENCES:
- [Background] Trupin L, Earnest G, San Pedro M, Balmes JR, Eisner MD, Yelin E, Katz PP, Blanc PD. The occupational burden of chronic obstructive pulmonary disease. Eur Respir J. 2003 Sep;22(3):462-9. doi: 10.1183/09031936.03.00094203. PMID 14516136
- [Background] Blanc PD, Eisner MD, Trupin L, Yelin EH, Katz PP, Balmes JR. The association between occupational factors and adverse health outcomes in chronic obstructive pulmonary disease. Occup Environ Med. 2004 Aug;61(8):661-7. doi: 10.1136/oem.2003.010058. PMID 15258271